CLINICAL TRIAL: NCT01456208
Title: Vascular Disease and Hbp: Pai-1, Insulin and Genes (Crc): Hypertension Phenotype
Brief Title: Genetic Mechanisms in Human Hypertension
Status: Terminated | Type: Observational
Why Stopped: Funding stopped
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gordon H. Williams, MD, Chief, Cardiovascular Endocrinology Section, Brigham and Women's Hospital
Other Study IDs: 1999P002189
Record Dates: First submitted 2011-09-28; First posted 2011-10-20 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — p-Aminohippuric Acid; Angiotensin II; Norepinephrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — urine, blood, DNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Para-aminohippuric Acid — Aminohippurate sodium is an agent to measure effective renal plasma flow (ERPF). It is the sodium salt of para-aminohippuric acid, commonly abbreviated "PAH".
  Other Names: PAH
Drug: Angiotensin II — Angiotensin II (Ang II) is a naturally occurring hormone whose primary purpose is to regulate the body's internal volume. It accomplishes this task by influencing the function of a variety of organs and tissues. It increases aldosterone secretion from the adrenal gland. It causes blood vessels to contract, particularly renal blood vessels, and it modifies the way the heart works.
  Other Names: AngII; AII
Drug: Norepinephrine — A hormone that is normally present in your body, which regulates your blood pressure.
  Other Names: NE

SUMMARY:
Thank you for your interest in the investigators Genetics and Blood Pressure Research Study. The National Institutes of Health are sponsoring us to investigate why patients develop high blood pressure, atherosclerosis (hardening of the arteries), and heart disease. There are two parts of the investigators research program. The first part is a screening visit. At this visit you will be given a brief physical exam and will be asked questions concerning your medical history. During the same visit you will have your blood drawn for routine screening and to prepare DNA for genetic testing. You will also be asked to collect a urine sample for routine screening.

If the doctor finds that you are a healthy candidate you will be invited to participate in the second part of the study. During Phase II, the investigators will perform physiological tests after you are placed on a low salt diet and again after you are placed on a high salt diet. If you are on blood pressure medication, it may be necessary to discontinue taking your present medication for up to three months before beginning the study. Patients discontinuing their current blood pressure medication may be placed on a different blood pressure medication during this washout period if necessary to maintain blood pressure at pre-study levels. The investigators will take you off all medications at about two weeks prior to your scheduled in-patient study (overnight visits).

Once your blood pressure medications are discontinued, you will be closely monitored to make sure you do not encounter any difficulty. If you do not own a home blood pressure monitor, the investigators will provide one for you to use during the study so that you can keep a daily record of your blood pressure readings. The investigators will ask you to call us every three days to report your blood pressure readings. Less than 20% of patients have any significant increase in their blood pressure during this short time off of therapy. After you have stopped taking your medication, dieticians at the hospital will make you low salt meals to eat at home for seven days. On the seventh day of the low salt diet, you will be asked to begin a 24-hour urine collection that you will bring with you when you are admitted to the hospital that evening. That morning, you will be required to come to the Clinical Research Center for a one-hour test to check if your body is in the correct salt balance. You will return that evening to the inpatient Clinical Research Center where you will be admitted for your study that will occur the next morning. On the morning of your low salt study, you will have naturally occurring hormones administered and blood samples drawn from an intravenous needle. The investigators will also take ultrasound pictures of your heart to see how salt and hormones affect the way the heart functions. These tests will last approximately five hours and you will be discharged around 2:00 PM. For the next five days, you will be placed on a high salt diet. During these five days, you will eat all your own food, but the investigators will give you some supplements to eat with your meals. After five days on your high salt diet, on the morning of your second admission to the hospital, you will be asked to begin a final 24-hour urine collection. That morning, you will again be required to come to the Clinical Research Center for a one-hour test to check if your body is in the correct salt balance. You will return that evening to the inpatient Clinical Research Center where you will be admitted for your final study that will occur the next morning. The same study that was done for the low salt study will be repeated for the high salt study. You will be discharged around 2:00 p.m. This study will determine if you are salt-sensitive. In addition, the investigators hope to learn more about the hormones that regulate your blood pressure and the genes responsible for regulating those hormones.

You will be placed back on your initial blood pressure medication (if you are on any) and returned to your regular physician for care. The investigators will provide clinically relevant information to you and your physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* A history of hypertension diagnosis and/or use of hypertension medications
* BMI < or equal to 40

Exclusion Criteria:

* Any other major illnesses
* Subjects with current excessive alcohol use (greater than 12 oz/ETOH/week) or recreational drug use
* BMI > 40
* Taking birth control or contraceptive hormone shots or implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age 18-65
  * A history of hypertension diagnosis and/or use of hypertension medications
  * BMI < or equal to 40
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 1999-10; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Independent Genetic Variants in the R-A-A System Predict Characteristics of Specific Intermediate Phenotypes of Hypertension (non-modulation and low renin). | 13 years
  1. Frequency of AGT minor allele homozygotics in non-modulating hypertension.
  2. Frequency of ALAP minor allele homozygotics in non-modulating hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon H Williams, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States